CLINICAL TRIAL: NCT07139574
Title: Impact of Music Therapy on Labor Pain and Anxiety: A Randomized Controlled Trial in Tunisian Women
Brief Title: Music Therapy for Labor Pain and Anxiety
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Tunis El Manar (Other)
Responsible Party: Principal Investigator, Nesrine Souayeh, Associate Professor, University Tunis El Manar
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 03/2025
Record Dates: First submitted 2025-08-17; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Labor Pain; Anxiety
Keywords: music therapy; anxiety; pain management; labor; randomized controlled trial
MeSH Terms: conditions — Labor Pain; Anxiety Disorders; Agnosia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music group (Experimental): The intervention consists of music therapy administered during the latent and active phases of labor. Music is delivered through headphones or speakers and includes slow, instrumental, non-lyrical tracks (60-80 beats per minute), selected in collaboration with the participant. The intervention is applied for a minimum duration of 30 minutes and follows established clinical guidelines for therapeutic music use. Standard monitoring of maternal and fetal well-being is maintained throughout the intervention.
  Interventions: Other: Music Therapy During Labor
- Control Group (No Intervention): This group received routine care during labor (monitoring of labor progression, vital signs, and fetal heart rate monitoring).
  No specific pain management techniques were used for this group.

INTERVENTIONS:
Other: Music Therapy During Labor — This intervention involves the use of patient-selected, slow-tempo (60-80 bpm), non-lyrical instrumental music administered via headphones or speakers during the latent and active phases of labor. The music selection is guided to ensure therapeutic suitability (e.g., calming rhythm, absence of lyrics) and is delivered for a minimum of 30 minutes. The intervention is non-pharmacological, individualized, and adheres to WHO and clinical music therapy recommendations. It is distinguished by its personalized music choice, delivery timing, and structured application within labor progression monitoring.
  Arms: Music group

SUMMARY:
This multicenter randomized controlled trial evaluates the effectiveness of music therapy in reducing pain and anxiety during the latent and active phases of labor in Tunisian women. Participants are randomized to receive either music therapy or standard care. Primary outcomes are pain (VAS) and anxiety (STAI-Y). Secondary outcomes include labor duration, maternal and fetal vital signs, neonatal outcomes, and maternal satisfaction.

DETAILED DESCRIPTION:
This study investigates the impact of music therapy on pain and anxiety management during labor in Tunisian parturients. Given the limited access to pharmacological analgesia in many public maternity units, the trial explores music as a non-pharmacological, low-cost, and patient-centered intervention. Eligible women in labor are randomly assigned to either a music therapy group or a control group receiving standard care. Music is administered during the latent and active phases following established clinical guidelines (slow tempo, non-lyrical, patient-guided selection). The study evaluates changes in pain intensity, anxiety levels, labor progression, maternal-fetal physiological parameters, neonatal outcomes, and maternal satisfaction. Findings aim to inform labor care practices and promote integrative approaches in resource-limited settings.

ELIGIBILITY:
Inclusion Criteria:

* Married Tunisian women with a singleton, low-risk pregnancy.
* Admitted in the latent phase of spontaneous labor, as diagnosed by a midwife or resident.
* Planned vaginal delivery.
* Parity < 4.
* Gestational age between 37 and 41 weeks of amenorrhea.
* Attended at least 4 prenatal consultations.
* Normal physical and mental health status.
* No known fetal anomalies.
* Estimated fetal weight between 2500-4000 g.
* Cephalic presentation.
* Normal fetal heart rate and uterine contraction tracings.
* Able to read, write, and understand study-related information.
* Provided written informed consent.

Exclusion Criteria:

* Women who received epidural analgesia during labor.
* Presence of auricular malformations.
* Difficulty in understanding or completing the VAS or STAI-Y assessments.
* Serious medical or psychiatric disorders.
* Multiple gestation or pregnancies requiring immediate intervention.
* Preterm (<37 weeks) or post-term (>41 weeks) pregnancies.
* Premature rupture of membranes.
* Clinical chorioamnionitis or other infections (including HIV).
* History of severe obstetric complications (e.g., cephalopelvic disproportion, intrauterine fetal death )

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Pain level | 30 minutes after completing the music session
  Pain intensity will be measured using a 10-cm Visual Analogue Scale (VAS), ranging from 0 = no pain to 10 = worst imaginable pain.
Anxiety level | 30 minutes after completing the music session
  Anxiety level will be measured using the State-Trait Anxiety Inventory, Form Y (STAI-Y), with higher scores indicating greater anxiety.

SECONDARY OUTCOMES:
Maternal pulse rate | 30 minutes after completing the music session
  Maternal pulse rate will be maesured in beat per minute 30 mn after listening to the musioc selection
Maternal arterial pressure | 30 minutes after completing the music session
  Maternal arterial pressure will be maesured in mmHg
Apgar score | 5 minutes after delivery
  the foetal pgar score was maesures on a scale from 0 to 10 five minutes after delivery
Maternal satisfaction | 2 hours after delivery
  Maternal satisfaction was maesured by a likert scale from 1 to 10 2 hours after delivery

CONTACTS AND LOCATIONS:
Locations (1):
- Ben Arous regional Hospital, Ben Arous, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data (IPD) will not be shared because of concerns regarding patient confidentiality and the absence of institutional infrastructure for secure data sharing.

REFERENCES:
- [Background] Vaid R, Fareed A, Farhat S, Hammoud Z, Asif MI, Ochani S, Jaber MH. Sounds of comfort: the impact of music therapy on labor pain and anxiety in primigravida women during vaginal delivery: a systematic review and meta-analysis. Reprod Health. 2025 May 9;22(1):67. doi: 10.1186/s12978-025-02023-z. PMID 40346658
- [Background] Santivanez-Acosta R, Tapia-Lopez ELN, Santero M. Music Therapy in Pain and Anxiety Management during Labor: A Systematic Review and Meta-Analysis. Medicina (Kaunas). 2020 Oct 10;56(10):526. doi: 10.3390/medicina56100526. PMID 33050409
- [Background] Guo H, Que M, Shen J, Nie Q, Chen Y, Huang Q, Jin A. Effect of Music Therapy Combined with Free Position Delivery on Labor Pain and Birth Outcomes. Appl Bionics Biomech. 2022 May 11;2022:8963656. doi: 10.1155/2022/8963656. eCollection 2022. PMID 35600844